CLINICAL TRIAL: NCT04125498
Title: The S-CARE Trial: Manual Treatment for C-sections Scars, a Pilot Study.
Acronym: S-CARE
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment during pandemic was impossible to achieve
Sponsor: Studio Osteopatico Busto Arsizio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S-Care pilot
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2021-03

CONDITIONS: Cesarean Section Complications; Cesarean Section; Complications, Wound, Infection (Following Delivery)
Keywords: adhesions; cicatrix; c-section; scar; manual treatment
MeSH Terms: conditions — Wounds and Injuries; Infections; Tissue Adhesions; Cicatrix | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: randomized triple-blinded
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The gynecologist, the radiologist and the statistician will be blinded to group allocation.
  Participants will have similar manual treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- OMT (Active Comparator): Osteopathic manual treatment
  Interventions: Other: Osteopathic treatment
- OMT plus self-massage (Active Comparator): Patients will be submitted to OMT and then they will be invited to practice a self-massage at home.
  Interventions: Other: Osteopathic treatment; Other: Self-massage
- Placebo (Sham Comparator): Similar to OMT without pressure.
  Interventions: Other: Placebo treatment
- Placebo plus self-massage (Active Comparator): Patients will be submitted to placebo manual treatment and then they will be invited to practice a self-massage at home.
  Interventions: Other: Placebo treatment; Other: Self-massage

INTERVENTIONS:
Other: Osteopathic treatment — Manual treatment that aims to release myofascial tensions
  Arms: OMT; OMT plus self-massage
Other: Placebo treatment — Similar to OMT without pressure
  Arms: Placebo; Placebo plus self-massage
Other: Self-massage — Women will be instructed to perform self-massage at home once a day for 5 minutes.
  Arms: OMT plus self-massage; Placebo plus self-massage

SUMMARY:
This study aims to examine the effects of an osteopathic treatment on adhesions related to c-sections scars.

DETAILED DESCRIPTION:
The rates of caesarean sections are growing throughout the world, with recent rates (in 2016) in Europe of 25%, in North America of 32.3% and in South America of 40.5%.

The incidence of intra-abdominal adhesions in women undergoing to repeated caesarean sections is constantly increasing.

Labor and surgical time are significantly longer in patients with adhesions compared to patients without adhesions.

Furthermore, it has been estimated that about 10% of patients undergoing cesarean section experience chronic pain.

Despite of the big impact on the quality of life of patients and high cost for public health, treatments for adhesions are mostly surgical.

The identification of non-surgical treatments that aim to reduce cicatricial adhesions' formation is essential to decrease hospitalization times and associated complications.

The purpose of this study is to evaluate the effects of osteopathic treatment and self-massage on scars in women who underwent to a cesarean section. The main aim is to assess whether there is a change in the number, size and vascularization of of cesarean section adhesionsthrough Superb Microvascular Imaging (SMI).

ELIGIBILITY:
Inclusion Criteria:

* primiparous or multipara who have undergone a cesarean section with a completely healed scar will be included.
* women who had first menstruation after childbirth
* Women with or without pain or symptoms related to scarring or the presence of isthmocele will be included.

Exclusion Criteria:

* caesarean section performed in a period less than 6 months and over 3 years
* uterine prolapse
* scar treatments already performed (both manual and medical)
* absence of scar adhesions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women underwent to a c-section
Enrollment: 50 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Adhesions' number, size and vascularization | Changes from Baseline Adhesions' number, size and vascularization at 2 weeks and one month
  Evaluate through superb microvascular imaging. Correlation between adhesions and type/number of c-section
Adverse event | Number of adverse event occurred at one month
  Number and type of adverse events
Uterine niches | Changes in dimension of uterine niches at one month
  Evaluation of the presence and dimensions of uterine niches

SECONDARY OUTCOMES:
Reliability of osteopathic palpation through a questionnaire | At one week, two week and one month
  Comparison between osteopathic palpation and ultrasound results in the detection of adhesions
Inter-reliability of ultrasound evaluation | At one week, two week and one month
  Ultrasound results comparison between gynecologist and radiologist using a vascularization scale (grade from 0 to 4)
Self-massage compliance | At one month
  Questionnaire
Symptoms related to scar | At one week, two week and one month

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Lavazza, MSc, Principal Investigator — Studio Osteopatico Busto Arsizio
Locations (1):
- Studio Osteopatico Busto Arsizio, Busto Arsizio, Varese, Italy

IPD SHARING:
Plan to Share IPD: No